CLINICAL TRIAL: NCT04260464
Title: A PHASE 1, NON-RANDOMIZED, OPEN LABEL, SINGLE DOSE STUDY TO EVALUATE THE PHARMACOKINETICS, SAFETY AND TOLERABILITY OF PF-06700841 IN PARTICIPANTS WITH RENAL IMPAIRMENT AND IN HEALTHY PARTICIPANTS WITH NORMAL RENAL FUNCTION
Brief Title: Renal Impairment Study of PF-06700841
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: B7931048
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Results first posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteer; Renal Impairment
Keywords: Pharmacokinetics
MeSH Terms: conditions — Renal Insufficiency | interventions — PF-06700841

STUDY DESIGN:
Intervention Model Description: Single group
Masking Description: No Masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PF-06700841 Severe Renal Impairment (Experimental): This arm includes participants with severe renal impairment who will receive a single oral dose of 30 mg PF-06700841 on Day 1
  Interventions: Drug: PF-06700841
- PF-06700841 Normal Renal Function (Experimental): This arm includes participants with normal renal function who will receive a single oral dose of 30 mg PF-06700841 on Day 1
  Interventions: Drug: PF-06700841
- PF-06700841 Moderate Renal Impairment (Experimental): This arm includes participants with moderate renal impairment who will receive a single oral dose of 30 mg PF-06700841 on Day 1
  Interventions: Drug: PF-06700841
- PF-06700841 Mild Renal Impairment (Experimental): This arm includes participants with mild renal impairment who will receive a single oral dose of 30 mg PF-06700841 on Day 1
  Interventions: Drug: PF-06700841

INTERVENTIONS:
Drug: PF-06700841 — A single dose of 30 mg PF-06700841 will be administered on Day 1

SUMMARY:
The purpose of this study is to characterize the effect of kidney impairment on the blood concentrations of PF-06700841 and its major metabolite. Findings from this study will be used to develop dosing recommendations so that the dose and/or dosing interval may be adjusted appropriately in the presence of kidney disease.

DETAILED DESCRIPTION:
This is a Phase 1 non-randomized, open-label, parallel cohort, multi-site study to investigate the effect of renal impairment on the pharmacokinetics, safety and tolerability of PF-06700841 after a single oral dose of 30 mg. Subjects will be selected and categorized into normal renal function or renal impairment groups based on their estimated glomerular filtration rate. Part 1: A total of approximately 16 subjects will be enrolled; approximately 8 subjects with severe renal impairment and approximately 8 with normal renal function. After statistical evaluation of results from Part 1, Part 2 may be conducted with approximately 8 subjects each with moderate and mild renal impairment. The total duration of participation from Screening visit to Day 4 will be a maximum of 32 days and from Screening visit to Follow-up/Contact Visit will a maximum of 67 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants who are between the ages of 18 and 75 years, inclusive, at the Screening visit.
* Body mass index (BMI) of ≥17.5 to ≤40 kg/m2; and a total body weight >50 kg.
* Normal, Severe, Moderate and Mild renal function at 2 Screening visits.
* Stable drug regimen

Exclusion Criteria:

* Renal transplant recipients.
* Urinary incontinence without catheterization.
* Subjects with clinically significant infections within the past 6 months prior to first dose of study drug, evidence of active or chronic infection requiring oral treatment within 4 weeks prior to first dose
* Known history of pulmonary embolism or recurrent deep vein thrombosis
* Any condition possibly affecting drug absorption (eg, prior bariatric surgery, gastrectomy, ileal resection).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Investigational Drug Services (IDS) University of Miami Hospitals and Clinics, Research Pharmacy, Miami, Florida
  - University of Miami Division of Clinical Pharmacology, Miami, Florida
  - Prism Research LLC dba Nucleus Network, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7931048

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adult participants with normal renal function and adult participants with renal impairment were enrolled in this study.
Pre-assignment Details: A total of 30 participants who met the eligibility criteria were assigned and treated.
Groups:
- Severe Renal Impairment: Participants with estimated glomerular filtration rate (eGFR) <30 ml/min and not requiring dialysis were categorized into the severe renal impairment arm. Participants received a single dose of PF-06700841 30 mg tablets (2 tablets as 1 x 5 mg and 1 x 25 mg) orally.
- Normal Renal Function: Participants with eGFR ≥90 mL/min were categorized into the normal renal function arm. Participants received a single dose of PF-06700841 30 mg tablets (2 tablets as 1 × 5 mg and 1 × 25 mg) orally.
- Moderate Renal Impairment: Participants with eGFR ≥30 to <60 mL/min were categorized into the moderate renal impairment arm. Participants received a single dose of PF-06700841 30 mg tablets (2 tablets as 1 × 5 mg and 1 × 25 mg) orally.
- Mild Renal Impairment: Participants with eGFR ≥60 to <89 mL/min were categorized into the mild renal impairment arm. Participants received a single dose of PF-06700841 30 mg tablets (2 tablets as 1 × 5 mg and 1 × 25 mg) orally.
Period: Overall Study
Arm/Group | Severe Renal Impairment | Normal Renal Function | Moderate Renal Impairment | Mild Renal Impairment
Started | 8 | 7 | 7 | 8
Completed | 8 | 7 | 7 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who were assigned to investigational product and took at least 1 dose of investigational product.
Groups:
- Severe Renal Impairment: Participants with eGFR <30 ml/min and not requiring dialysis were categorized into the severe renal impairment arm. Participants received a single dose of PF-06700841 30 mg tablets (2 tablets as 1 x 5 mg and 1 x 25 mg) orally.
- Total: Total of all reporting groups
Arm/Group | Severe Renal Impairment | Normal Renal Function | Moderate Renal Impairment | Mild Renal Impairment | Total
Number analyzed (Participants) | 8 | 7 | 7 | 8 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Mean (SD) | 65.9 (7.57) | 62.4 (5.38) | 68.4 (4.24) | 61.5 (6.16) | 64.5 (6.36)
Age, Customized [Number; unit: Participants]
  45-64 Years | 3 | 6 | 1 | 6 | 16
  >=65 Years | 5 | 1 | 6 | 2 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 4 | 8
  Male | 7 | 6 | 5 | 4 | 22
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 8 | 5 | 6 | 8 | 27
  Black or African American | 0 | 2 | 1 | 0 | 3
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 4 | 4 | 2 | 4 | 14
  Not Hispanic or Latino | 4 | 3 | 5 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-06700841 Following Single Oral Dose Administration in Participants With Renal Impairment and in Healthy Participants With Normal Renal Function
Description: Cmax is the maximum observed plasma concentration of PF-06700841 within 72 hours post dose, which was observed directly from the plasma concentration-time data.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hours after dose
Population: The PK concentration population is defined as all participants assigned to investigational product and treated who have at least 1 concentration measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Severe Renal Impairment | Normal Renal Function | Moderate Renal Impairment | Mild Renal Impairment
Number analyzed (Participants) | 8 | 7 | 7 | 8
ng/mL | 303.2 (34) | 275.2 (27) | 341.8 (17) | 260.3 (89)
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Normal Renal Function; Analysis of variance (ANOVA) was used to compare the natural log transformed Cmax for PF-06700841 between the normal renal function group (Reference) and the severe impaired renal function group (Test). Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% confidence intervals (CIs) were obtained from the model; Test type: Other; Test/Reference Ratio = 110.15, 95% CI 2-sided [83.76 to 144.86]
Statistical Analysis 2: Comparison: Normal Renal Function vs Mild Renal Impairment; ANOVA was used to compare the natural log transformed Cmax for PF-06700841 between the normal renal function group (Reference) and the mild impaired renal function group (Test). Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% confidence intervals (CIs) were obtained from the model; Test type: Other; Test/Reference Ratio = 94.58, 90% CI 2-sided [55.84 to 160.19]
Statistical Analysis 3: Comparison: Normal Renal Function vs Moderate Renal Impairment; ANOVA was used to compare the natural log transformed Cmax for PF-06700841 between the normal renal function group (Reference) and the moderate impaired renal function group (Test). Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% confidence intervals (CIs) were obtained from the model; Test type: Other; Test/Reference Ratio = 124.20, 90% CI 2-sided [100.24 to 153.89]

2. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to Infinity (AUCinf) of PF-06700841 Following Single Oral Dose Administration in Participants With Renal Impairment and in Healthy Participants With Normal Renal Function
Description: AUCinf was area under the concentration-time curve from time 0 to infinity, which was calculated for PF-06700841 from the concentration-time data.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hours after dose
Population: The PK parameter analysis population is defined as all participants assigned to investigational product and treated who have at least 1 of the PK parameters of primary interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Severe Renal Impairment | Normal Renal Function | Moderate Renal Impairment | Mild Renal Impairment
Number analyzed (Participants) | 8 | 6 | 7 | 8
ng*hr/mL | 2013 (57) | 1796 (77) | 2652 (75) | 1274 (199)
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Normal Renal Function; ANOVA was used to compare the natural log transformed AUCinf for PF-06700841 between normal renal function group (Reference) and the severe impaired renal function group (Test). Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs were obtained from the model; Test type: Other; Test/Reference Ratio = 112.08, 95% CI 2-sided [60.85 to 206.45]
Statistical Analysis 2: Comparison: Normal Renal Function vs Mild Renal Impairment; ANOVA was used to compare the natural log transformed AUCinf for PF-06700841 between normal renal function group (Reference) and the mild impaired renal function group (Test). Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs were obtained from the model; Test type: Other; Test/Reference Ratio = 70.97, 90% CI 2-sided [27.60 to 182.49]
Statistical Analysis 3: Comparison: Normal Renal Function vs Moderate Renal Impairment; ANOVA was used to compare the natural log transformed AUCinf for PF-06700841 between normal renal function group (Reference) and the moderate impaired renal function group (Test). Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs were obtained from the model; Test type: Other; Test/Reference Ratio = 147.70, 90% CI 2-sided [75.17 to 290.21]

3. Primary Outcome: Cmax of PF-06802530 (M1) Following Single Oral Dose Administration in Participants With Renal Impairment and in Healthy Participants With Normal Renal Function
Description: Cmax is the maximum observed plasma concentration of PF-06802530 (M1), a major metabolite of PF-06700841 within 72 hours post dose, which was observed directly from the plasma concentration-time data.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hours after dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Severe Renal Impairment | Normal Renal Function | Moderate Renal Impairment | Mild Renal Impairment
Number analyzed (Participants) | 8 | 7 | 7 | 8
ng/mL | 250.4 (26) | 141.0 (32) | 172.1 (46) | 187.1 (43)
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Normal Renal Function; ANOVA was used to compare the natural log transformed Cmax for M1 between normal renal function group (Reference) and the severe impaired renal function group (Test). Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs were obtained from the model; Test type: Other; Test/Reference Ratio = 177.53, 95% CI 2-sided [135.82 to 232.04]
Statistical Analysis 2: Comparison: Normal Renal Function vs Mild Renal Impairment; ANOVA was used to compare the natural log transformed Cmax for M1 between normal renal function group (Reference) and the mild impaired renal function group (Test). Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs were obtained from the model; Test type: Other; Test/Reference Ratio = 132.69, 90% CI 2-sided [95.08 to 185.17]
Statistical Analysis 3: Comparison: Normal Renal Function vs Moderate Renal Impairment; ANOVA was used to compare the natural log transformed Cmax for M1 between normal renal function group (Reference) and the moderate impaired renal function group (Test). Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs were obtained from the model; Test type: Other; Test/Reference Ratio = 122.04, 90% CI 2-sided [84.47 to 176.30]

4. Primary Outcome: AUCinf of PF-06802530 (M1) Following Single Oral Dose Administration in Participants With Renal Impairment and in Healthy Participants With Normal Renal Function
Description: AUCinf was area under the concentration-time curve from time 0 to infinity, which was calculated for PF-06802530 (M1), a major metabolite of PF-06700841 from the concentration-time data.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hours after dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Severe Renal Impairment | Normal Renal Function | Moderate Renal Impairment | Mild Renal Impairment
Number analyzed (Participants) | 7 | 7 | 7 | 8
ng*hr/mL | 7756 (41) | 1739 (24) | 3984 (15) | 2515 (32)
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Normal Renal Function; ANOVA was used to compare the natural log transformed AUCinf for M1 between normal renal function group (Reference) and the severe impaired renal function group (Test). Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs were obtained from the model; Test type: Other; Test/Reference Ratio = 445.99, 95% CI 2-sided [326.55 to 609.13]
Statistical Analysis 2: Comparison: Normal Renal Function vs Mild Renal Impairment; ANOVA was used to compare the natural log transformed AUCinf for M1 between normal renal function group (Reference) and the mild impaired renal function group (Test). Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs were obtained from the model; Test type: Other; Test/Reference Ratio = 144.63, 90% CI 2-sided [112.76 to 185.50]
Statistical Analysis 3: Comparison: Normal Renal Function vs Moderate Renal Impairment; ANOVA was used to compare the natural log transformed AUCinf for M1 between normal renal function group (Reference) and the moderate impaired renal function group (Test). Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs were obtained from the model; Test type: Other; Test/Reference Ratio = 229.12, 90% CI 2-sided [189.97 to 276.35]

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Any events occurring following start of treatment or increasing in severity after the start of the treatment were counted as treatment emergent. An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect. Severe adverse events is an event that prevents normal everyday activities which is a category utilized for rating the intensity of an event.
Time Frame: From screening (Day-28 to Day -2) to up to 35 days after the study treatment (for a period of up to 63 days)
Population: The analysis population included all assigned to investigational product and who take at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Renal Impairment | Normal Renal Function | Moderate Renal Impairment | Mild Renal Impairment
Number analyzed (Participants) | 8 | 7 | 7 | 8
Participants
  Participants with adverse events | 2 | 0 | 1 | 3
  Participants with serious adverse events | 0 | 0 | 0 | 0
  Participants with severe adverse events | 0 | 0 | 0 | 0
  Participants discontinued from study due to adverse events | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities Without Regard to Baseline Abnormality
Description: The hematology, clinical chemistry and urinalysis abnormalities were summarized in accordance with the sponsor reporting standards without regard to baseline abnormality. Baseline is defined as the last planned predose measurement taken on Day -1.
Time Frame: Baseline (Day -1) and Day 4
Population: The analysis population included all participants assigned to investigational product and who take at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Renal Impairment | Normal Renal Function | Moderate Renal Impairment | Mild Renal Impairment
Number analyzed (Participants) | 8 | 7 | 7 | 8
Participants
  Hematology-Hemoglobin (HGB) (g/dL) <0.8✕lower limit of normal (LLN) | 2 | 0 | 0 | 0
  Hematology-Hematocrit (%) <0.8✕LLN | 1 | 0 | 0 | 0
  Hematology-Erythrocytes (10^6/mm^3) <0.8✕LLN | 1 | 0 | 0 | 0
  Hematology- Erythromycin (Ery.) Mean Corpuscular HGB (pg/cell) >1.1✕upper limit of normal (ULN) | 1 | 0 | 0 | 0
  Hematology-Ery. Mean Corpuscular HGB Concentration (g/dL) <0.9✕LLN | 0 | 0 | 1 | 0
  Hematology-Lymphocytes/Leukocytes (%) <0.8✕LLN | 1 | 0 | 1 | 0
  Hematology-Lymphocytes/Leukocytes (%) >1.2✕ULN | 0 | 1 | 0 | 0
  Hematology-Eosinophils/Leukocytes (%) >1.2✕ULN | 2 | 0 | 0 | 0
  Clinical chemistry-Blood Urea Nitrogen (mg/dL) >1.3✕ULN | 8 | 0 | 2 | 0
  Clinical chemistry-Creatinine (mg/dL) >1.3✕ULN | 8 | 0 | 1 | 0
  Clinical chemistry-Urate (mg/dL) > 1.2✕ULN | 5 | 0 | 0 | 1
  Clinical chemistry-Potassium (mEq/L) >1.1✕ULN | 0 | 0 | 0 | 1
  Clinical chemistry-Bicarbonate (mEq/L) <0.9✕LLN | 1 | 0 | 0 | 0
  Clinical chemistry-Glucose (mg/dL) >1.5✕ULN | 1 | 0 | 4 | 2
  Urinalysis-Urine Glucose ≥1 | 2 | 0 | 1 | 1
  Urinalysis-Urine Protein ≥1 | 2 | 0 | 0 | 0
  Urinalysis-Urine Hemoglobin ≥1 | 0 | 0 | 0 | 1
  Urinalysis-Urine Leukocyte Esterase ≥1 | 1 | 1 | 0 | 2

7. Secondary Outcome: Number of Participants With Post-baseline Vital Sign Abnormalities
Description: Vital Signs were assessed against the criteria specified in the sponsor reporting standards for potential clinical concerns. Vital sign abnormalities criteria included: 1) Systolic blood pressure (BP) in millimeters of mercury (mmHg): <90 mmHg with increase or decrease from baseline of ≥30 mmHg with high and low post baseline values; 2) Diastolic blood pressure (BP) (mmHg): <50 mmHg with increase or decrease from baseline of ≥20 mmHg with high and low post baseline values; 3) Supine pulse rate in beats per minutes (bpm): >120 or <40 bpm. Categories with at least 1 participant having vital sign abnormality in any of the reporting arms, were reported in this outcome measure. Baseline is defined as the last planned predose measurement taken on Day 1.
Time Frame: Baseline (Day 1) and Day 4
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Renal Impairment | Normal Renal Function | Moderate Renal Impairment | Mild Renal Impairment
Number analyzed (Participants) | 8 | 7 | 7 | 8
Participants | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Post-baseline Electrocardiogram (ECG) Abnormalities
Description: ECG abnormalities criteria included: 1) QTc interval adjusted according to Bazett formula (QTcB) in millisecond (msec): > 450, >480, >500, increase from baseline >30, increase from baseline >60; 2) QTc interval adjusted according to Fridericia formula (QTcF) (msec): >450, >480, >500, increase from baseline >30, increase from baseline >60. Categories with at least 1 participant having ECG abnormality in any of the reporting arms, were reported in this outcome measure. Baseline is defined as the last planned predose measurement taken on Day 1.
Time Frame: 0 hr pre-dose and 1-, 3-, and 6-hours post-dose on Day 1; Day 4
Population: All assigned to investigational product and who take at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Renal Impairment | Normal Renal Function | Moderate Renal Impairment | Mild Renal Impairment
Number analyzed (Participants) | 8 | 7 | 7 | 8
Participants
  QTcB interval, single beat (msec): 450 < Value ≤ 480 | 2 | 0 | 1 | 3
  QTcB interval, single beat (msec): 30 ≤ Change ≤ 60 | 0 | 0 | 0 | 3
  QTcF interval, single beat (msec): 450 < Value ≤ 480 | 2 | 1 | 1 | 0
  QTcF interval, single beat (msec): 30 ≤ Change ≤ 60 | 0 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: From screening (Day-28 to Day -2) to up to 35 days after the study treatment (for a period of up to 63 days)
Arm/Group | Severe Renal Impairment | Normal Renal Function | Moderate Renal Impairment | Mild Renal Impairment
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 2/8 | 0/7 | 1/7 | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Severe Renal Impairment (N=8) | Normal Renal Function (N=7) | Moderate Renal Impairment (N=7) | Mild Renal Impairment (N=8)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-11-20): https://cdn.clinicaltrials.gov/large-docs/64/NCT04260464/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT04260464/SAP_001.pdf